CLINICAL TRIAL: NCT05663619
Title: The Effect of Virtual Reality Distraction on Anxiety Level During Dental Treatment Among Anxious Pediatric Patients: A Randomized Clinical Trial
Brief Title: Virtual Reality Distraction and Dental Anxiety Among Anxious Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Osama M Felemban, Associate Professor in Pediatric Dentistry, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAUFD20221207
Record Dates: First submitted 2022-12-07; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Children's Dental Anxiety
Keywords: Dental anxiety; heart rate; salivary cortisol; virtual reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality distraction (VRD) (Experimental): In the VRD group, participants wore a VRD device and watched a previously selected favorite cartoon during the prophylactic dental treatment.
  Interventions: Device: Virtual Reality Distraction during dental treatment of children.
- control group (Active Comparator): In the control group, participants received their treatment while watching a previously selected favorite cartoon on a regular screen.
  Interventions: Other: Control: watching cartoon on screen as distraction during dental treatment of children.

INTERVENTIONS:
Device: Virtual Reality Distraction during dental treatment of children. — One of the behavior management techniques used with children in dental clinics to allow for delivering quality dental treatment is the use of Virtual Reality distraction (VRD). Virtual reality distraction immerses the patient in an environment generated by a computer and works by simulating as many senses as possible: vision, hearing, and touch. In dentistry, VRD has exhibited great results in reducing anxiety and fear among children and adolescents compared to those who received no intervention or more conventional BMTs. VRD may allow the dentist to provide more efficient dental treatments, ranging from simple anesthesia to more advanced forms of dental treatment
  Arms: Virtual Reality distraction (VRD)
Other: Control: watching cartoon on screen as distraction during dental treatment of children. — The American Academy of Pediatric Dentistry (AAPD) recommends a series of non-pharmacological behavior management techniques for managing children during dental care including distraction. Distraction is defined by AAPD as "the technique of diverting the patient's attention from what may be perceived as an unpleasant procedure". It is widely used as it provides an effective and relaxing experience during treatment.
  Arms: control group

SUMMARY:
Objective: This study evaluated the effect of Virtual Reality Distraction (VRD) on dental anxiety among anxious children undergoing prophylactic dental treatment by utilizing both subjective (Venham Anxiety and Behavioral Rating Scale (VABRS)) and objective (heart rate (HR) and salivary cortisol level (SCL)) measures. Method and Materials: This randomized controlled study included 36 6- to 14-year-old healthy and anxious children who needed prophylactic dental treatment and who had a history of previous dental treatment. The eligible children's anxiety level was evaluated using a modified version of Abeer Dental Anxiety Scale-Arabic version (M-ACDAS) and those who scored at least 14 or more out of 21 were included. Participants were randomly distributed to either the VRD or control group. In the VRD group, participants wore the VRD device during prophylactic dental treatment. In the control group, subjects received their treatment while watching a video cartoon on a regular screen. The participants were videotaped during the treatment and their HR was recorded at four time points. Also, a sample from each participant's saliva was collected twice, at the baseline and after the procedure.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of virtual reality distraction among 6- to 14-year-old anxious children undergoing prophylactic dental treatment by utilizing both subjective (Venham Anxiety and Behavioral Rating Scale (VABRS)) and objective (heart rate and salivary cortisol level) measures.

This two-arms parallel randomized controlled study was conducted at the Department of Pediatric Dentistry at King Abdulaziz University Dental Hospital (KAUDH) between January and May 2022, after obtaining the ethical approval from the Research Ethics Committee of the Faculty of Dentistry (341-11-21) at King Abdulaziz University. The study is reported according to the protocol established by the Consolidated Standards of Reporting Trials (CONSORT) statement (18).

The inclusion criteria were 6- to 14-year-old, healthy children with a history of previous dental treatment. The included subjects also had to have high dental anxiety (high score on a modified version of Abeer Children Dental Anxiety Scale (M-ACDAS)) . Children with visual or auditory deficits, a history of epilepsy, and/or anxiety disorder, and non-Arabic speaking children were excluded.

Records of pediatric patients on the dental treatment waiting list were reviewed and potentially eligible children were contacted via the phone. The aim of the study was introduced to the parents/guardians, and upon agreement to participate, an appointment was scheduled.

Abeer Children Dental Anxiety Scale (ACDAS), a cognitive dental anxiety scale, is the first Arabic validated cognitive dental anxiety scale developed to measure anxiety in children and adolescents. It consists of 19 self-reported questions arranged in a logical order to assess dental anxiety in children (19). In this study, the ACDAS was modified (M-ACDAS), and only seven of the 19 self-reported questions were included to avoid a lengthy questionnaire with the children (Figure 1). Each question can be scored 1, 2, or 3 by choosing between three faces with different expressions. The first face is a smily face and reflects the feeling of being relaxed, happy, and not scared, while the second face represents a neutral feeling; and the third face is a sad face and represents anxious and scared feeling. The children were asked to circle the face that best represented his/her response to the question. Therefore, the total values ranged from 7 to 21. The M-ACDAS was used at the beginning of the scheduled appointment in the waiting area to assess the pre-treatment anxiety level of the potentially eligible children. Those who scored 14 (66.7% of the maximum score) or more were considered anxious and were included in the study. Those who scored less than 14 in the M-ACDAS were excluded from the study.

An Arabic consent form was obtained from the parents/guardians, and a verbal assent was obtained from the child before participation. The participants' age, gender, the timing, type of treatment provided, and behavior during their most recent dental visit were also recorded.

A stratified block randomization process was used to randomize the 36 participants into either a VRD or a control group. The participants were stratified by gender and then a block size of six was used in each stratum. The sequence of assignments in each block was generated using a random number generator. To ensure allocation concealment, the allocation assignment and sequence were kept with a dental assistant not involved in the study. In the VRD group, participants wore a VRD device and watched a previously selected favorite cartoon during the prophylactic dental treatment. The device was introduced to the participants using the Tell-Show-Do technique at the beginning of the appointment. In the control group, participants received their treatment while watching a previously selected favorite cartoon on a regular screen. For both groups, only speakers with no headphones were used.

The subjects underwent a dental prophylactic treatment performed by a single trained dental intern using a low-speed handpiece and a rubber cup with prophy paste. The dental treatment was conducted in the same order, the upper right, upper left, lower left, and lower right quadrants with all the participants. The participants were allowed to choose the prophy paste flavor (Bubble Gum, Cherry Tart, Concord grape, Mint Parfait, Raspberry Jam, and Valencia Orange). During the treatment, the HR was recorded using a pulse oximeter (TECNO-GAS pulse oximeter VITAL TEST) at four-time points: (1) in the waiting area as a baseline; (2) in the dental chair before starting the procedure and after the VRD device or the regular screen were turned on; (3) during prophylactic dental treatment (after prophy of the two quadrants in the upper arch was completed); (4) after the procedure was completed and before taking off the VRD device in the VRD group or turning off the regular screen in the control group.

During the treatment, participants were videotaped using a high-resolution camera. Later, two trained and calibrated evaluators assessed the participant's anxiety using the VABRS independently. The scale consists of five defined behavioral categories ranging from zero to five. A higher score indicates a greater level of anxiety (20).

Two saliva samples were collected from each participant: (1) as a baseline in the waiting area; (2) after the dental procedure was completed. Approximately two mL of saliva was collected using Salivettes®, and the samples were stored at -20oC until evaluation. To minimize the effects of the diurnal cortisol cycle, all study procedures and saliva sample collection were performed between 10:00 am and 2:00 pm. The cortisol levels were measured using the Cortisol Saliva Enzyme-Linked Immunosorbent Assay (ELISA) Assay Kit (ab 154996- cortisol ELISA kit, Abcam, UK) following the manufacturer's instructions.

Sample size and statistical analysis A sample size of 18 in each group will have 80% power to detect a difference in means of -1.5 assuming that the common standard deviation is 1.5 with a 5% two-sided significance level. The Statistical Package for Social Science software for Windows was used for the statistical analysis (SPSS, Chicago, IL, USA). The participants' baseline characteristics were compared using the Mann-Whitney U test, chi-square test, or Fisher exact test. The Mann-Whitney U test was used to compare the three outcomes of the research (HR, SCL, and VABRS) between the VRD and control groups. The significance threshold was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 6- to 14-year-old.
* Healthy.
* With a history of previous dental treatment.
* High dental anxiety (high score on a modified version of Abeer Children Dental Anxiety Scale (M-ACDAS)).

Exclusion Criteria:

* Visual or auditory deficits.
* History of epilepsy, and/or anxiety disorder.
* Non-Arabic speaking children.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Heart rate | (1) as a baseline in the waiting area before dental treatment; (2) in the dental chair immediately before starting the procedure; (3) during prophylactic dental treatment procedure; (4) immediately after the procedure was completed
  The HR was recorded using a pulse oximeter
Venham Anxiety and Behavioral Rating Scale | 1 day (during dental treatment procedure)
  During the treatment, participants were videotaped using a high-resolution camera. Later, two trained and calibrated evaluators assessed the participant's anxiety using the Venham Anxiety and Behavioral Rating Scale independently. The scale consists of five defined behavioral categories ranging from zero to five. A higher score indicates a greater level of anxiety.
Change in Salivary cortisol levels. | (1) as a baseline in the waiting area before dental treatment; (2) immediately after the dental procedure was completed
  Two saliva samples were collected from each participant: (1) as a baseline in the waiting area; (2) after the dental procedure was completed. Approximately two mL of saliva was collected using Salivettes®, and the samples were stored at -20oC until evaluation. To minimize the effects of the diurnal cortisol cycle, all study procedures and saliva sample collection were performed between 10:00 am and 2:00 pm. The cortisol levels were measured using the Cortisol Saliva Enzyme-Linked Immunosorbent Assay (ELISA) Assay Kit (ab 154996- cortisol ELISA kit, Abcam, UK) following the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
There is no intent to share IPD with other researchers.

REFERENCES:
- [Background] Felemban OM, Alshamrani RM, Aljeddawi DH, Bagher SM. Effect of virtual reality distraction on pain and anxiety during infiltration anesthesia in pediatric patients: a randomized clinical trial. BMC Oral Health. 2021 Jun 25;21(1):321. doi: 10.1186/s12903-021-01678-x. PMID 34172032
- [Background] Shetty V, Suresh LR, Hegde AM. Effect of Virtual Reality Distraction on Pain and Anxiety During Dental Treatment in 5 to 8 Year Old Children. J Clin Pediatr Dent. 2019;43(2):97-102. doi: 10.17796/1053-4625-43.2.5. Epub 2019 Feb 7. PMID 30730798
- [Background] Rao DG, Havale R, Nagaraj M, Karobari NM, Latha AM, Tharay N, Shrutha SP. Assessment of Efficacy of Virtual Reality Distraction in Reducing Pain Perception and Anxiety in Children Aged 6-10 Years: A Behavioral Interventional Study. Int J Clin Pediatr Dent. 2019 Nov-Dec;12(6):510-513. doi: 10.5005/jp-journals-10005-1694. PMID 32440065